CLINICAL TRIAL: NCT04869722
Title: Modifying Whey Protein Fortified Drinks and Foods to Improve Perception, Whilst Accounting for Individual Differences in Age (At Home Study)
Brief Title: Modifying Whey Protein Fortified Drinks and Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Volac International Limited (Unknown)
Responsible Party: Principal Investigator, Lisa Methven, Professor in Food and Sensory Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 20/35
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Individual Difference; Food Sensitivity; Food Preferences
Keywords: Older adults; Mouthdrying; Protein fortified foods and beverages
MeSH Terms: conditions — Food Intolerance; Food Preferences

STUDY DESIGN:
Intervention Model Description: This study involves both a crossover design where each participant tastes different protein fortified products with an appropriate break between the tasting. It is also both a within and between groups design as the responses from the older volunteers will be compared with the younger volunteers. The study will be conducted single blind as it not feasible to blind the researcher. Each participant will attend 1 study visits and all products will be presented with random blinding codes.
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid Model (Experimental): Whey protein beverages varying in protein levels
  Interventions: Behavioral: Liquid Model
- Solid Model (Experimental): Protein fortified scones varying in fat levels
  Interventions: Behavioral: Solid Model

INTERVENTIONS:
Behavioral: Liquid Model — Whey protein beverages will be used, with the amount of protein varied to study the effect on perception of the products (using sensory methods rating mouthdrying and discrimination tests 'which sample is more mouthdrying') all measured at home.
  Arms: Liquid Model
Behavioral: Solid Model — Protein fortified scones will be used, with the amount of fat varied to study the effect on perception of the products (using sensory methods rating mouthdrying and discrimination tests 'which sample is more mouthdrying') all measured at home.
  Arms: Solid Model

SUMMARY:
This study aims to investigate whether consumers differ in mouthdrying sensitivity and if mouthdrying can be modulated.

DETAILED DESCRIPTION:
1. To investigate whether older adults are more sensitive to whey protein derived mouthdrying compared with younger adults
2. To investigate whether increasing fat levels in a solid whey protein model influences mouthdrying perception

ELIGIBILITY:
Inclusion Criteria:

* Age (18-30 years or over 65 years)
* Healthy

Exclusion Criteria:

* Relevant food allergies or intolerance
* Outside age criteria
* Diabetic
* Had oral surgery
* Had a stroke
* Smoker
* Cancer Taking prescribed medication that could influence study outcomes Anyone who currently has COVID-19 symptoms or who has had COVID-19 within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Whey Protein Beverages Mouthdrying Just Noticeable Difference Threshold | 1 hour (sampled at visit one)
  Perceived mouthdrying from whey protein beverages varying in protein levels using data from sensory methods (discrimination tests asking "which sample is more mouthdrying" in each pair)

SECONDARY OUTCOMES:
Whey Protein Beverages Mouthdrying Ratings | 1 hour (sampled at visit one)
  Perceived mouthdrying from whey protein beverages varying in protein levels using data from sensory methods (rating mouthdrying)
Modulating mouthdrying | 1 hour (sampled at visit one)
  Perceived mouthdrying from protein fortified scones varying in fat levels using data from sensory methods (rating mouthdrying as well as discrimination tests "which sample is more mouthdrying")

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Science, University of Reading, Reading, Berkshire, United Kingdom, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Norton V, Lignou S, Bull SP, Gosney MA, Methven L. An Investigation of the Influence of Age and Saliva Flow on the Oral Retention of Whey Protein and Its Potential Effect on the Perception and Acceptance of Whey Protein Beverages. Nutrients. 2020 Aug 19;12(9):2506. doi: 10.3390/nu12092506. PMID 32825104
- [Background] Norton V, Lignou S, Bull SP, Gosney MA, Methven L. Consistent Effects of Whey Protein Fortification on Consumer Perception and Liking of Solid Food Matrices (Cakes and Biscuits) Regardless of Age and Saliva Flow. Foods. 2020 Sep 21;9(9):1328. doi: 10.3390/foods9091328. PMID 32967299
- [Background] Bull SP, Hong Y, Khutoryanskiy VV, Parker JK, Faka M, Methven L. Whey protein mouth drying influenced by thermal denaturation. Food Qual Prefer. 2017 Mar;56(Pt B):233-240. doi: 10.1016/j.foodqual.2016.03.008. PMID 28260840
- [Background] Withers CA, Lewis MJ, Gosney MA, Methven L. Potential sources of mouth drying in beverages fortified with dairy proteins: A comparison of casein- and whey-rich ingredients. J Dairy Sci. 2014 Mar;97(3):1233-47. doi: 10.3168/jds.2013-7273. Epub 2014 Jan 17. PMID 24440265